CLINICAL TRIAL: NCT02792998
Title: A 2-Stage Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IW-1701 Tablets in Healthy Subjects in a Double-blind, Placebo-controlled, Multiple-ascending-dose Stage and an Open-label, Single-dose, Crossover Food-effect Stage
Brief Title: A Trial of IW-1701, A Stimulator of Soluble Guanylate Cyclase (sGC), in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-1701-102
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- IW-1701 (Experimental): IW-1701 tablets administered orally in multiple ascending dose.
  Interventions: Drug: IW-1701
- Placebo (Placebo Comparator): Matching placebo tablets administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IW-1701 — IW-1701 Tablet
  Arms: IW-1701
Drug: Placebo — Matching Placebo Tablet
  Arms: Placebo

SUMMARY:
The objectives of this study are:

Stage 1: To assess the safety, tolerability, pharmacokinetic (PK) profile and pharmacodynamic (PD) effects of a range of doses of IW-1701 tablets administered orally to healthy subjects over 7 days of repeated dosing

Stage 2: To assess the safety, tolerability, PK profile and PD effects of IW-1701 tablets administered orally to healthy subjects, in fed and fasted states, in an open-label, single-dose, 2-period, 2-sequence crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an ambulatory male or female between 18 and 55 years old at the screening visit
* Subject's body mass index score is > 18.5 and < 30.0 kg/m2 at the screening visit
* Women of childbearing potential must have a negative pregnancy test at the time of check-in and must agree to use double-barrier contraception throughout the duration of the study
* Subject is in good health and has no clinically significant findings on a physical examination
* Other inclusion criteria per protocol

Exclusion Criteria:

* History of any clinically significant medical conditions
* Other exclusion criteria per protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Event | 47 Days
Maximum observed plasma concentration [Cmax] | 47 Days
  Maximum observed Plasma Concentration
Area under the plasma concentration time curve during a dosing interval [AUC] | 47 Days
  Area under the plasma concentration time curve during a dosing interval
Time of maximum observed plasma concentration [Tmax] | 47 Days
  Time of maximum observed plasma concentration
Blood Pressure | 47 Days

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Early Phase Unit, San Antonio, Texas, United States